CLINICAL TRIAL: NCT05029323
Title: Validation of a Novel Simplified Head up Tilt Test (HUTT) Protocol Versus the Conventional Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Vincenzo Russo, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 22062020
Record Dates: First submitted 2021-07-27; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Syncope; Syncope;Heat Induced
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional HUTT (Active Comparator): All patients with unexplained syncope at initial evaluation with indication to perform a Head up tilt test (HUTT) randomized to "conventional" HUTT protocol characterized by a stabilization phase of 5 min in the supine position; a passive phase of 10 min at a tilt angle of 60 degrees; aprovocation phase of further 10 min after 300 micrograms NTG sublingual spray.
  Interventions: Diagnostic Test: Conventional HUTT
- Fast HUTT (Experimental): All patients with unexplained syncope at initial evaluation with indication to perform a Head up tilt test (HUTT) randomized to "fast" HUTT protocol characterized by a stabilization phase of 5 min in the supine position; a passive phase of 10 min at a tilt angle of 60 degrees; a provocation phase of further 10 min after 300 micrograms NTG sublingual spray.
  Interventions: Diagnostic Test: Fast HUTT

INTERVENTIONS:
Diagnostic Test: Fast HUTT — Fast HUTT protocol stabilization phase of 5 min in the supine position; passive phase of 10 min at a tilt angle of 60 degrees; provocation phase of further 10 min after 300 micrograms NTG sublingual spray.
  Arms: Fast HUTT
Diagnostic Test: Conventional HUTT — Conventional HUTT protocol stabilization phase of 5 min in the supine position; passive phase of 20 min at a tilt angle of 60 degrees; provocation phase of further 15 min after 300 micrograms NTG sublingual spray.
  Arms: Conventional HUTT

SUMMARY:
The purpose of the study is to compare the positivity rate associated with a novel simplified Tilt-Table (TT) test protocol versus the conventional TT protocol

DETAILED DESCRIPTION:
All patients with unexplained syncope at initial evaluation with indication to perform a Head up tilt test (HUTT) will be randomized to "conventional" HUTT protocol or "fast" HUTT protocol characterized by a stabilization phase of 5 min in the supine position; a passive phase of 10 min at a tilt angle of 60 degrees; a provocation phase of further 10 min after 300 micrograms NTG sublingual spray. The novel simplified "fast" HUTT protocol has been designed to provide non inferior positivity rates as compared with the conventional protocol in the selected population.

ELIGIBILITY:
Inclusion Criteria:

* All patients with unexplained syncope at initial evaluation and indication to perform HUTT

Exclusion Criteria:

* No informed consent
* PM/ICD device recipients

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-01-07 (Estimated); Study Completion 2023-01-07 (Estimated)

PRIMARY OUTCOMES:
HUTT positivity rate during passive phase | through study completion, an average of 1 year
  The study endpoint is the number of patients who experienced syncope during the passive phase of HUTT.
HUTT positivity rate during active phase | through study completion, an average of 1 year
  The study endpoint is the number of patients who experienced syncope during the active phase of HUTT.

SECONDARY OUTCOMES:
The type of HUTT-induced syncope during passive phase | through study completion, an average of 1 year
  The secondary study endpoint is the number of patients with cardioinhibitory HUTT-syncope during the passive phase of HUTT.
The type of HUTT-induced syncope during active phase | through study completion, an average of 1 year
  The secondary study endpoint is the number of patients with cardioinhibitory HUTT-syncope during the active phase of HUTT.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russo, MD PhD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: No